CLINICAL TRIAL: NCT05397782
Title: Pilot Study: Effects of Flourish Vaginal Care System in Women With Recurrent Symptomatic Urinary Tract Infections
Brief Title: Effects of Flourish on Recurrent Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vaginal Biome Science (Other)
Collaborators: Urology Associates, P.C., Tennessee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: rUTI0522
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Urinary Tract Infections
Keywords: vaginal microbiome; microbiome; probiotic; lactobacillus; vulvovaginal symptoms questionnaire; vaginal pH
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: A single group of women with recurrent symptomatic UTI will be studied longitudinally while using the intervention system. Results will be compared with historical controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pilot Group: Flourish HEC (Experimental): All women in the study will use the Flourish HEC Vaginal Care System for 6 months. Flourish HEC consists of 3 products: 1) Balance, an external feminine wash; 2) BioNourish, a vaginal moisturizing gel; and 3) BiopHresh, a homeopathic vaginal suppository with probiotics. Products are pH-balanced to match healthy vaginal pH (3.5-4.5). BioNourish is formulated to be iso-osmotic with vaginal fluid. Balance and BioNourish contain lactic acid. BiopHresh contains 7 strains of lactobacilli, including Lactobacillus crispatus and other species found in healthy vaginas or shown to be effective probiotics strains.
  Interventions: Device: BioNourish, a component of Flourish HEC

INTERVENTIONS:
Device: BioNourish, a component of Flourish HEC — BioNourish, one of three parts of the Flourish HEC system, is a vaginal moisturizing gel - a Class II medical device with FDA 510k clearance obtained in 2020.

SUMMARY:
An over-the-counter vaginal care system is being tested to see if it may be effective in preventing recurrence of symptomatic urinary tract infection (UTI) in women who have had multiple UTIs within the past year.

DETAILED DESCRIPTION:
Women who have a urinary tract infection (UTI) may experience a recurrence within weeks or months of treatment. Some women may experience 8 or more UTIs in a single year, leading to multiple rounds of antibiotics, with the individual risks to organs and risk of antibiotic resistance growing with each round. Alternative methods for prevention of recurrent UTI is therefore desirable. This study will test whether women who use a commercially available, over-the-counter vaginal care system may be able to reduce recurrences of UTI over a six-month period. This is a pilot study designed to determine whether a larger randomized controlled trial in the future would be justified.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal cis women aged 18-52 who are in generally good health
2. History of at least 2 UTIs in the past six months, or three prior UTIs in the past year, documented in the medical record. At least one must be culture-proven.

Exclusion Criteria:

1. Pregnant or trying to become pregnant
2. Lactating
3. Immunosuppressed
4. Known allergies to aloe vera or to other components of Restore®, Balance or BiopHresh®
5. Known vaginal infection other than BV or yeast infection at time of screening
6. Women who have needed changes to medical intervention or in-office procedures in the last 3 months
7. Women using vaginal acidifying agents or spermicides for contraception
8. Women who wear a pessary

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Vaginal Microbiome | Baseline to 3 months
  The vaginal microbiome will be assessed using next-generation sequencing (NGS) technology to assign the biome to one of 5 "community state types" (CST). The outcome will examine whether the vaginal microbiome changes from an unhealthy one (IV or III) to a healthy one (I, II, or V).
Vaginal Microbiome | Baseline to 6 months
  The vaginal microbiome will be assessed using next-generation sequencing (NGS) technology to assign the biome to one of 5 "community state types" (CST). The outcome will examine whether the vaginal microbiome changes from an unhealthy one (IV or III) to a healthy one (I, II, or V).
Vaginal Microbiome | 3 months to 6 months
  The vaginal microbiome will be assessed using next-generation sequencing (NGS) technology to assign the biome to one of 5 "community state types" (CST). The outcome will examine whether the vaginal microbiome changes from an unhealthy one (IV or III) to a healthy one (I, II, or V).
UTI recurrence | Baseline to 6 months
  Frequency of symptomatic UTI over study duration will be assessed (number of occurrences per person). UTI will be diagnosed when one or more symptoms is present (urinary urgency, frequency, sense of burning, pelvic pain, fever, flank pain) along with one or more confirming lab tests (positive culture, urine nitrites or leukocytes).

SECONDARY OUTCOMES:
Associations between microbes and UTI | Baseline to 6 months.
  Using the NGS sequencing data from primary outcomes 1, 2, and 3, statistical modeling will be used to determine if the presence of specific individual bacteria or combinations of two or more species are associated with increased frequency of UTI.
Vaginal pH | Baseline to 6 months
  Vaginal pH will be tested by pH strip.
Vaginal pH | Baseline to 3 months
  Vaginal pH will be tested by pH strip.
Vaginal pH | 3 months to 6 months
  Vaginal pH will be tested by pH strip.
Vulvovaginal symptoms questionnaire (VSQ) + addendum | Baseline
  Vulvovaginal symptoms will be assessed by questionnaire. Both the validated VSQ and additional questions not previously validated will be used. Most questions will be asked using a 4-point Likert scale (0=not at all, 4 = all the time), except those which are binary in nature.
Vulvovaginal symptoms questionnaire (VSQ) + addendum | 3 months
  Vulvovaginal symptoms will be assessed by questionnaire. Both the validated VSQ and additional questions not previously validated will be used. Most questions will be asked using a 4-point Likert scale (0=not at all, 4 = all the time), except those which are binary in nature.
Vulvovaginal symptoms questionnaire (VSQ) + addendum | 6 months
  Vulvovaginal symptoms will be assessed by questionnaire. Both the validated VSQ and additional questions not previously validated will be used. Most questions will be asked using a 4-point Likert scale (0=not at all, 4 = all the time), except those which are binary in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Faught, DNP, Principal Investigator — Women's Institute of Sexual Health / Urology Associates
Locations (1):
- WISH A Place for Women, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No